CLINICAL TRIAL: NCT04101500
Title: Clinical Study on the Efficacy of Compound Sodium Chlorate and Aminophylline Tablets for Mild to Moderate Acute Exacerbation of Chronic Obstructive Pulmonary Disease(COPD).
Brief Title: Effect of Compound Sodium Chlorate and Aminophylline Tablets on Chronic Obstructive Pulmonary Disease(COPD).
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Yang Jin, Department of Respiratory and Critical Care Medicine, NHC Key Laboratory of Pulmonary Diseases, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2018S446-1
Record Dates: First submitted 2019-09-18; First posted 2019-09-24 (Actual); Last update posted 2019-09-24 (Actual); Status verified 2019-09

CONDITIONS: Acute Exacerbation of Chronic Obstructive Pulmonary Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AECOPD(P+C1) (Placebo Comparator): Placebo Tablets(P) three times a day, one tablet at a time; combined with Compound Ipratropium Bromide Solution(C1) 2.5ml atomized inhalation twice a day.
  Interventions: Drug: Compound Ipratropium Bromide Solution(C1) for Inhalation; Drug: Placebo Tablets
- AECOPD(C1+C2) (Experimental): Compound Sodium Chlolate and Aminophylline Tablets(C2) three times a day, one tablet at a time; combined with Compound Ipratropium Bromide Solution(C1) 2.5ml atomized inhalation twice a day.
  Interventions: Drug: Compound Ipratropium Bromide Solution(C1) for Inhalation; Drug: Compound Sodium Chlolate and Aminophylline Tablets(C2)

INTERVENTIONS:
Drug: Compound Ipratropium Bromide Solution(C1) for Inhalation — The patient's condition and basic condition were the same in the experimental group and the control group.
  Other Names: CIBS(C1)
Drug: Compound Sodium Chlolate and Aminophylline Tablets(C2) — Applied only to the experimental group.
  Other Names: CSCAT(C2)
  Arms: AECOPD(C1+C2)
Drug: Placebo Tablets — Applied only to the control group.
  Other Names: PT
  Arms: AECOPD(P+C1)

SUMMARY:
Acute exacerbation of chronic obstructive pulmonary disease (AECOPD) is an important event in the management of chronic obstructive pulmonary disease. Compound sodium chlolate and aminophylline tablets are one of the most widely used drugs for the treatment of bronchial asthma and chronic bronchitis.

DETAILED DESCRIPTION:
Acute exacerbation of chronic obstructive pulmonary disease (AECOPD) is an unignorable event in the management of chronic obstructive pulmonary disease. It is crucial to seek for effective management strategy. Compound sodium chlolate and aminophylline tablets are one of the most widely used drugs for the treatment of bronchial asthma and chronic bronchitis. Compared with the local bronchodilator recommended by the guidelines, it has the advantages of convenient use and good patient compliance. For the purpose of optimize the management of acute exacerbation of chronic obstructive pulmonary disease and provide more convenient options, we compared the efficacy of combined compound sodium chlolate and aminophylline tablets with nebulized ipratropium bromide inhalation plus systemic glucocorticoids in the treatment of chronic obstructive pulmonary disease ranging from moderate degree to severe degree. We hope this research would benefit patients with chronic obstructive pulmonary, especially those in the grassroots.

ELIGIBILITY:
Inclusion Criteria:

- (1)All subjects must sign an informed consent form before participating in the clinical trial.

(2)Clinical diagnosis of AECOPD. (3)Must be able to swallow tablets.

Exclusion Criteria:

* (1)Heart disease. (2)Insulin dependent diabetes. (3)Tumor disease. (4)Thyroid disease. (5)Infectious diseases such as hepatitis B, active tuberculosis, etc. (6)Active peptic ulcer. (7)Allergic to related treatments. (8)Participate in other clinical trials within three months. (9)Women who are breast-feeding, pregnant or preparing for pregnancy.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
COPD assessment test(CAT) score | The above test was given to the experimental group and the control group on the first, fourth, and eighth days after the treatment.
  Observe the changes in the symptoms of dyspnea each time.The CAT score consists of eight items, each of which has options of 0, 1, 2, 3, 4, and 5. The lower the total score plus the score for the eight items, the lighter the symptoms of COPD.The first item, whether there is cough; the second item, sputum condition; the third item, whether there is chest tightness; the fourth item, when climbing a hill or climbing a layer of stairs, is there any breathlessness;the fifth item, whether chronic obstructive pulmonary disease affects housework; the sixth item, whether it affects going out; the seventh item, sleep situation; the eighth item, whether the energy is sufficient.
Potential of Hydrogen(PH),Partial pressure of oxygen(PO2),Partial pressure of carbon dioxide(PCO2) | The above test was given to the experimental group and the control group on the first, fourth, and eighth days after the treatment.
  Arterial blood gas values were monitored, the values measured at each examination were recorded, and changes between each time were observed.

SECONDARY OUTCOMES:
Forced Expiratory Volume in the first second (FEV1)/Forced Vital Capacity(FVC) | The above test was given to the test group and the control group on the first and eighth days after the treatment.
  Observe the changes in lung function each time.

CONTACTS AND LOCATIONS:
Overall Officials: Yang Jin, Principal Investigator — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China